CLINICAL TRIAL: NCT02391324
Title: Evaluation of the Effectiveness of Robotic Gait Training and Gait-focused Physical Therapy Programs for Children and Youth With Cerebral Palsy: A Mixed Methods Randomized Controlled Trial
Brief Title: Effectiveness of Robotic Gait Training and Physical Therapy for Children and Youth With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Holland Bloorview Kids Rehabilitation Hospital (Other); Shirley Ryan AbilityLab (Other); Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: RES0022460
Record Dates: First submitted 2015-03-06; First posted 2015-03-18 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lokomat (LOK) (Experimental): Two 50-minute sessions per week. The manualized LOK walking protocol provides methods for progressing/tracking including a 5-minute overground walking session after the LOK to facilitate transfer of motor learning from the LOK to usual walking devices. The goal-based LOK program uses a standardized approach to progressing LOK body weight and guidance support and includes upper body activities while walking to encourage dual tasking and improved posture, and motor imagery practice.
  Interventions: Procedure: Lokomat (LOK)
- Gait focused physical therapy (fPT) (Experimental): Two 50-minute sessions per week. Each weekly fPT session consists of 50 minutes of active treatment, a 'dose' equivalent to time spent in active treatment in the LOK arm. Techniques that focus on body structure changes will be not be permitted (e.g., inhibitive casting, kinesiotaping, functional electrical stimulation).
  Interventions: Procedure: Gait focused physical therapy (fPT)
- LOK + fPT (Experimental): Two 50-minute sessions per week. Children will receive both the LOK and the fPT protocols (content as described above for each) for the duration of the 8 to 10 week intervention phase. These will be given as two sessions of LOK one week alternating with two sessions of fPT the next week. The fPT will build on motor learning principles because the activities will allow the child to practice motor skills in a variety of different activities. Techniques focusing on body structure changes will be prohibited.
  Interventions: Procedure: LOK + fPT
- Maintenance therapy (No Intervention): Consists of maintenance therapy and a weekly email from the centre's research assistant to monitor any co-interventions. Maintenance may include range of motion/stretching and basic isometric strength home program as well as up to 10 minutes per day of exercise bicycle or treadmill or general walking practice.

INTERVENTIONS:
Procedure: Lokomat (LOK) — Physical therapy provided using a robotic gait training system (Lokomat).
  Other Names: Robotic Gait Training
  Arms: Lokomat (LOK)
Procedure: Gait focused physical therapy (fPT) — Overground physical therapy focussed on enhancing gait related motor skills
  Arms: Gait focused physical therapy (fPT)
Procedure: LOK + fPT — A combination of robotic gait training and gait focussed functional physical therapy.
  Arms: LOK + fPT

SUMMARY:
Robot assisted gait training is seen as a promising intervention for improving the walking abilities of children with cerebral palsy, but research to support its effectiveness compared to best practice physical therapy is lacking. This research consists of a randomized controlled trial (RCT) and a qualitative descriptive study that is linked with the RCT. The goal of the RCT is to compare: 1) a walking training program with the Lokomat® robotic device (LOK), 2) a functional physical therapy program (fPT) that includes activities to enhance balance/co-ordination/endurance and advanced motor skills conducted over 'real ground', 3) a combined Lokomat® + functional physical therapy (LOK+fPT) program, and 4) a regular maintenance therapy condition (CONT) for ambulatory children and youth with CP (aged 5- 18 years). The three intervention programs will consist of sixteen 50-minute sessions given twice weekly over 8 to 10 weeks. The primary objective of the RCT is to compare the four groups with respect to walking-related motor skills as measured by the Gross Motor Function Measure. The secondary objectives are to compare each intervention's impact on walking abilities, individualized goals, fitness, balance, physical activity levels, child's belief in ability to do physical activity, participation and quality of life. The investigators will also evaluate the extent of carryover or progress 3 months after the intervention. The qualitative part of the study will consist of interviews of children and parents after they have finished the study intervention. The information from the interviews will assist us with interpretation of the outcome results (areas of impact and amount of change) from the RCT. In particular, the interviews will 1) provide insight into their experiences with the trial interventions, 2) identify the mobility-related outcomes that are important to families and the factors that influence their preferences, and 3) explain the family values, experiences and contextual factors that influenced participation in the study. This research will provide information needed to allow clinicians and families to make informed choices about Lokomat therapy and physical therapy options in relation to their child's functional goals and abilities.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common cause of childhood physical disability, affecting 2.0-2.5 in 1000 children. CP represents a group of disorders of movement and posture with impairments (e.g., muscle weakness, decreased selective motor control, alterations in muscle tone, and impairment of postural control) that collectively affect functional mobility. About 65% of children/youth with CP use minimal or no assistive devices (leg braces, walkers, and/or wheelchairs) to walk (i.e., Gross Motor Function Classification System (GMFCS) Levels I and II) while children in GMFCS Levels III - V require varying degrees of bracing, walkers and other walking devices, wheelchairs, or assistance from others for mobility.

Robotic Assisted Gait training devices are increasingly used with children with CP to improve their gait related motor skills. The Lokomat® (LOK) is a commercially available robot assisted gait training system that uses robotics to simulate walking. It facilitates inter-limb co-ordination and gait cycle timing and provides variable degrees of body weight support and guidance.

This study represents the first adequately powered RCT to evaluate the effectiveness of robot assisted gait training for children with CP. The qualitative aspect will give contextual information to assist with interpretation of the RCT and provide valuable information about families' experiences with the interventions.

The research questions for this study are:

i) What is the comparative effectiveness of robot assisted gait training (LOK) and fPT program for improving gait related motor skills of ambulatory children and youth with CP? ii) Does combining LOK and fPT result in greater improvements in gait related motor skills of ambulatory children and youth with CP than robot assisted gait training or fPT alone? iii) What are families' experiences with trial participation and what implications do they have for interpretation of the quantitative results and the use of robot assisted gait training and fPT in clinical settings?

Methods This trial is a concurrent, mixed methods study. Specifically, the quantitative arm is a multi-centre RCT with four groups (22 factorial design, i.e., LOK absent/present, fPT absent/present) with two periods of post-intervention assessments (immediate and 3 months later). The RCT is linked with an interpretive descriptive qualitative study arm. The three study sites are Holland Bloorview (Toronto, Ontario, Canada), Glenrose Rehabilitation Hospital (Edmonton, Alberta, Canada) and Rehabilitation Institute of Chicago (Chicago, IL).

Participants - Children aged 5-18 with CP, GMFCS levels II and III. Inclusion/Exclusion criteria included in protocol in documents section.

Randomization - Following the baseline assessment, participants will be randomly allocated to one of the four groups using computer-generated random sequence.

Blinding Physical therapist assessors and data analysts will be blinded to group allocation.

TreatmentThere are three intervention groups: 1) LOK, 2) LOK + fPT, 3) fPT, and 4) one maintenance therapy control (CONT) arm. All three intervention groups will receive two 50-minute sessions per week, conducted over 8 -10 weeks. Children in all four groups can continue to participate in 'maintenance therapy'. Each child will be assigned to a treatment team of two trained PTs who will share responsibility for the 8 to 10 week intervention phase.

LOK - two 50-minute sessions on the Lokomat® per week. The study manualized LOK walking protocol provides methods for progressing/tracking including a 5-minute over ground walking session after the LOK to facilitate transfer of motor learning from the Lokomat to usual walking devices.

fPT Participants will Two 50-minute sessions per week. The manualized motor-learning based protocol forms the basis for this intervention. Its focus is on balance and multi-plane gait-based motor skills.

LOK + fPT group protocol: Participants will alternate between LOK and one fPT session per week for the duration of the 8 to 10 week intervention phase.

Monitoring co-interventionsMaintenance therapies such as home stretching and strengthening routines can be continued for all 4 groups throughout the study because these therapies have questionable efficacy, and will likely be equally used across all four groups as they are common PT recommendations.

Outcomes - All study outcomes will be measured pre-/post-intervention (< 10 days pre-intervention and post-completion), and at 3m follow-up (+/- 10 day window) by trained physical therapists. Data will be entered into REDCap.

Primary Outcome - The primary outcome measure is the Gross Motor Function Measure-66 (GMFM-66 Dimensions D (Stand) and E (Walk/Run/Jump).

Secondary Outcomes - Secondary outcomes are measures of walking capacity(6 minute walk test) fitness (adapted shuttle run test), balance (Pediatric Berg Balance Scale, Quality Function Measure (FM), and Activities Balance Confidence Scale), functional abilities (PEDI-CAT), physical activity levels (accelerometry), participation (Participation and Environment Measure for Children and Youth), physical activity self-efficacy (Self-Efficacy for Physical Activity), individualized goal attainment (Canadian Occupational Performance Measure (COPM) and Goal Attainment Scaling), and quality of life (KidScreen and Students' Life Satisfaction Scale).

Statistical Analysis - Data will be described (e.g., means, standard deviations, frequencies) for each intervention group and each stratification variable. Mixed-effects multiple linear regression models will be developed for each outcome with centre as a random effect, centre by intervention as an interaction (to assess centre effect), and other important variables (e.g., age and GMFCS level) as covariates. All main analyses will be based on intent-to-treat with secondary analyses of those with >80% adherence to their intervention.

Qualitative Component

The three objectives of the concurrent qualitative component are to explicate:

1. Child and parent experiences with the trial interventions and the values and previous experiences that shape their perceptions.
2. The mobility related outcomes that are important to families and factors that influence these views.
3. Child and family values, experiences and contextual factors that influenced participation in the trial, including the follow-up period.

Design Interpretive description

Sample selection- The investigators will invite a subset of child-parent dyads from each of the active interventions in the RCT. In addition, parents of children who were eligible but declined to participate in the RCT will be invited to participate in the qualitative component to address objective #3. The estimated sample size is (i.e., 6 child/parent dyads plus 3 parents from each site).

Data Collection - Parents will participate in 45-60 minute semi-structured, individual interviews conducted by one member of the research team. Participating parents of children in the RCT will be interviewed at 2 points within the trial: i) after completion of the COPM and prior to receiving the intervention, and ii) within one month of intervention completion.

Children from the RCT will participate in individual interviews at the end of their LOK/fPT intervention. A customizable "tool box" of age-appropriate child-friendly techniques including photographs and comic captioning, vignettes, and sentence starters will be used in a 30-45 minute semi-structured interview with the child without the parent present.

Data Management and Analysis Interviews will be digitally audio-recorded, transcribed verbatim by a professional transcriptionist, de-identified and imported into NVivo for data management. Two researchers will collaboratively identify general coding categories. The researchers will meet to establish consensus on the coding.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CP (any type), GMFCS Levels II and III
* Able to follow GMFM testing instructions, and to participate in a minimum of 30 minutes of active PT (as judged by the child's PT or physician if not followed by a PT)
* Able to reliably signal pain, fear and discomfort using verbal or nonverbal signals
* Passive range of motion (ROM) of hips and knees within minimum range requirement for LOK (hip and knee flexion contracture < 10 degrees, and knee valgus < 40 degrees).
* Parent/child agrees to attend 16 study intervention sessions (given within two 10-week periods), a LOK fitting/acclimatization session or fPT acclimatization session and the three assessment sessions during the course of the study.
* Parent agrees to contact of their primary PT (if not already involved by parent in the screening process) and their paediatrician or physiatrist to confirm eligibility.
* Parent agrees that regular PT (and other gross motor mobility therapies such as conductive education and MEDEK) will be discontinued from the time of the baseline assessment through the 8 to 10 weeks of the active intervention or control group. Note that home programs such as stretching and strengthening and treadmill and exercise bike riding (no more than 10 minutes total per day) will be permitted in all groups.

Exclusion Criteria:

* Botulinum Toxin injection within the past 4 months or planned within the next 6 months
* Fixed knee contracture > 10 degrees, knee valgus >40 degrees such that orthosis will not be adaptable to lower limbs.
* Hip instability/subluxation as demonstrated by a migration percentage > 45%
* Orthopaedic surgery (soft tissue releases) within the last 9 months, or lower limb bony surgery within the last 18 months
* Severe spasticity may be a contraindication as determined in Lokomat trial session using L-FORCE assessment.
* Any weightbearing restrictions.
* Seizure disorder unless fully controlled by medication and no evidence of seizure in the last 12 months and physician provides singed approval to enter the study
* Open skin lesions or vascular disorder of lower extremities
* Not able to co-operate or be positioned adequately within the LOK as shown during the fitting/acclimatisation session. -

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in gross motor abilities using the Gross Motor Function Measure (GMFM-66) from 0-8 and 0-20 weeks | Baseline, 8 weeks, 20 weeks
  A standardized measure of gross motor function for children with cerebral palsy

SECONDARY OUTCOMES:
Change in walking distance using the 6-Minute walk test from 0-8 and 0-20 weeks | Baseline, 8 weeks, 20 weeks
  Distance walked in 6 minutes
Change in individual goal attainment using the Canadian Occupational Performance Measure (COPM) performance ratings from 0-8 and 0-20 weeks | Baseline, 8 weeks, 20 weeks
  Individualized goal setting tool and outcome measure (ratings of performance and satisfaction with performance)
Change in individual goal attainment using Goal Attainment Scaling (GAS) from 0-8 and 0-20 weeks | Baseline, 8 weeks, 20 weeks
Change in anaerobic capacity using the Adapted Shuttle Run Test from 0-8 and 0-20 weeks | Baseline, 8 weeks, 20 weeks
Change in Pediatric Berg Balance Scale from 0-8 and 0-20 weeks | Baseline, 8 weeks, 20 weeks
Change in Quality FM from 0-8 and 0-20 weeks | Baseline, 8 weeks, 20 weeks
Change in confidence in performing ambulatory abilities as measured by the Activities Balance Confidence Scale from 0-8 and 0-20 weeks | Baseline, 8 weeks, 20 weeks
Change in functional abilities as measured by the PEDI-CAT from 0-8 and 0-20 weeks | Baseline, 8 weeks, 20 weeks
Change in # of steps/day from 0-8 and 0-20 weeks as measured with an accelerometer. | Baseline, 8 weeks, 20 weeks
Change in self-efficacy for physical activity as measured by the Physical Activity Self-efficacy scale | Baseline, 8 weeks, 20 weeks
  Change in Self-efficacy for Physical Activity score from 0-8 and 0-20 weeks
Change in the participation measured using the Participation and Environment Measure for Children and Youth (PEM-CY) from 0-8 and 0-20 weeks | Baseline, 8 weeks, 20 weeks
Change in quality of life using the Kidscreen from 0-8 and 0-20 weeks | Baseline, 8 weeks, 20 weeks-up
Change in quality of life using the Life Satisfaction Scale from 0-8 and 0-20 weeks | Baseline, 8 weeks, 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Wright, PhD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital; Lesley Wiart, PhD, Principal Investigator — University of Alberta
Locations (3):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Wiart L, Rosychuk RJ, Wright FV. Evaluation of the effectiveness of robotic gait training and gait-focused physical therapy programs for children and youth with cerebral palsy: a mixed methods RCT. BMC Neurol. 2016 Jun 2;16:86. doi: 10.1186/s12883-016-0582-7. PMID 27255908